CLINICAL TRIAL: NCT05690269
Title: Impact of Skin Pigmentation on Accuracy of Pulse Oximetry
Brief Title: Oximeters and Skin Pigment: Impact of Skin Pigmentation on Accuracy of Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dina Gomaa, Assistant Professor, University of Cincinnati
Other Study IDs: HRP-503
Record Dates: First submitted 2022-12-20; First posted 2023-01-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypoxemia; Hyperoxia; Pigment Skin
Keywords: SpO2, SaO2,Hypoxemia
MeSH Terms: conditions — Hypoxia; Hyperoxia; Pigmentation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: SpO2 and SaO2 comparison — Several pulse oximeter will be place on patients fingers a few minutes before arterial blood gases. SpO2 will be recorded during that time and up to 10 minutes.

SUMMARY:
Finger pulse oximetry SpO2 is widely used to estimate arterial oxygen saturation SaO2. Current Spo2 targets do not take into consideration the many variables that affect that correlation in particular skin pigmentation.

This study aims to evaluate different FDA approved pulse oximeters (Nonin co-pilot, massimo Radical 7, Philips-standard of care monitor, innovo premium iP900BP, nellcor PM1000N, Nano100) with SaO2 reference values obtained by an arterial blood gas in subjects with different skin pigments measured by a skin color scale as well as self-identification of race.

DETAILED DESCRIPTION:
The oximeters that will be evaluated are nonin co-pilot, massimo Radical 7, Philips (standard care), Innovo Premium iP900BP, nellcor PM1000N and USA medical supply Nano100. The sensors used will be reusable digital sensors for all oximeters. Oximeters will have been placed on patients' fingers (3 fingers on each hand) during an initial phase of clinical stability. Due to the impact of the fingers used for SpO2 measurement and bias that might be caused by right hand versus left hand, oximeters will be randomized to different fingers and hands for each patient. Measurements will be made when the SpO2 with the usual oximeter is <97% as recommended and in the absence of changes of the respiratory parameters in the last 10 minutes. A set of measures that will include all the oximeters tested will be used. Once the oximeters are installed, at least 2 minutes will run out to let the oximeters reach steady state. Then when a standard of care blood gas is obtained, measurements will be taken simultaneously to the drawing of a standard care arterial blood gas by a clinician in the ICU. While the clinician takes the arterial blood gas, a picture will be simultaneously taken of the SpO2 readings shown by each oximeter, in addition to taking vital signs, O2 flow or FiO2.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Patients admitted to the Intensive Care Unit
* Patient has arterial line

Exclusion Criteria:

* No signal with the oximeter
* Missing digits preventing application of all probes simultaneously
* No requirement for arterial blood gases
* Pigmented nails, fake nails, or nail polish
* Methemoglobinemia
* Patient in isolation (multi-resistant bacteria, C-Difficile, COVID-19)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Difference between SpO2 and the SaO2 value in all studied oximeters | At the time of arterial blood samples collection. Approximately 15 minutes.
  Difference between oximeter SpO2 and the corresponding SaO2 value

SECONDARY OUTCOMES:
Evaluation of oximeter accuracy in subpopulations of subjects with hypothermia | At the time of arterial blood samples collection. Approximately 15 minutes.
  Evaluation of oximeter accuracy in subpopulations of subjects with hypothermia (body temperature < 34 degrees C) and subjects requiring vasoactive infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Gomaa, MSc, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided